CLINICAL TRIAL: NCT00813150
Title: Randomized Phase III Study on Bortezomib and Low-Dose Dexamethasone With or Without Continuous Low-Dose Oral Cyclophosphamide for Primary Refractory or Relapsed Multiple Myeloma
Brief Title: Study of Bortezomib and Dexamethasone With or Without Cyclophosphamide in Patients With Relapsed or Not Controllable Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015247; 26866138MMY3022 (Other: Janssen-Cilag G.m.b.H, Germany); 2008-003213-27 (EudraCT Number)
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Bortezomib; Dexamethasone; Cyclophosphamide; Oncology
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Dexamethasone; Bortezomib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vd (bortezomib + dexamethasone) (Experimental): Participants received bortezomib at a dose of 1.3 mg/m² body surface area (BSA) for eight 3-week cycles. Within each cycle it was administered twice weekly (on Days 1, 4, 8, and 11) followed by a 10-day rest period (Days 12 through 21). They received single oral doses of 20 mg dexamethasone on Days
  1 and 2, 4 and 5, 8 and 9, and 11 and 12 of each cycle.
  Interventions: Drug: Dexamethasone; Drug: Bortezomib
- Vcd (bortezomib + low-dose dexamethasone + cyclophosphamide) (Active Comparator): Participants received bortezomib at a dose of 1.3 mg/m² body surface area (BSA) for eight 3-week cycles. Within each cycle it was administered twice weekly (on Days 1, 4, 8, and 11) followed by a 10-day rest period (Days 12 through 21). They received single oral doses of 20 mg dexamethasone on Days 1 and 2, 4 and 5, 8 and 9, and 11 and 12 of each cycle and single oral doses of 50 mg cyclophosphamide on a once daily basis from Day 1, Cycle 1 continuously until Day 21, Cycle 8.
  Interventions: Drug: Dexamethasone; Drug: Bortezomib; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Dexamethasone — Type=exact number, number=20, unit=mg, form=tablet, route=oral. The patients will receive 20 mg of dexamethasone on days 1+2,4+5,8+9,11+12 for 21 days for 8 cycles.
Drug: Bortezomib — Type=exact number, number=1.3, unit=mg, form=injection, route=intravenous. The patients will receive 1.3mg/m2 on days 1,4,8,11 for 21 days for 8 cycles.
Drug: Cyclophosphamide — Type=exact number, number=50, unit=mg, form=tablet, route=oral. The patients will receive 50 mg of cyclophosphamide once daily continuously from cycle 1 to 8.
  Arms: Vcd (bortezomib + low-dose dexamethasone + cyclophosphamide)

SUMMARY:
The purpose of this study is to compare bortezomib, dexamethasone and cyclophosphamide to bortezomib and dexamethasone alone for primary refractory or relapsed multiple myeloma.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, randomized (the study drug is assigned by chance), controlled, open-label (all people involved in the study know the identity of the assigned drug), parallel (each group of patients will be treated at the same time) group phase III study to determine the efficacy of the standard therapy of bortezomib and low dose dexamethasone in combination with or without continuous low dose oral cyclophosphamide for primary refractory or relapsed myeloma patients (1st - 3rd relapse). The study will consist of screening period, which may last from day -14 until day -1 before application of the first dose of bortezomib (on cycle 1, day 1), treatment phase begins on cycle 1 day 1 and continues until completion or discontinuation of all study drugs and follow-up phase. All patients will be followed up after end of treatment regardless of their response. Eligible patients will be randomized in 1:1 ratio to receive either treatment arms (Group A: receiving bortezomib plus dexamethasone or Group B receiving bortezomib plus dexamethasone plus cyclophosphamide). Patients will receive up to eight 3-weeks treatment cycles, unless they experience either unacceptable toxicity or if the patients request to withdraw from the study. The maximum number of cycles is dependent on patient response and investigator's discretion. It is recommended that patients with a confirmed complete response (CR) receive 2 additional cycles beyond a confirmation. Patients who do not achieve a CR but a partial response will receive a total of 8 cycles. For patients achieving stable disease it is within the investigator's discretion to continue study treatment beyond 6 cycles, after discussion with the sponsor. After completion of treatment the patients will be followed up every 12 weeks for up to 72 weeks. If the study is still ongoing a further follow up period will be done every 26 weeks until study end, or until the patient reaches progressive disease or start of alternative anti-myeloma therapy, if earlier. In case progressive disease (PD) has already been established during the treatment phase the patients will not enter the follow-up phase. In case of PD or start of alternative anti-myeloma treatment before the end of study the follow-up phase will be discontinued for the patient but the date of death of the patient will be documented (if applicable) before the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with multiple myeloma
* Primary refractory multiple myeloma or relapsed following 1 to 3 previous lines of therapy
* Karnofsky performance status must be equal to 60 percentage (ie, better or equal performance than requiring some help and taking care of most personal requirements)
* Has life expectancy estimated at screening must be of at least 6 months
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Not received more than three previous lines of therapy for multiple myeloma
* Not received nitrosoureas or any other chemotherapy or immunotherapy or antibody therapy for multiple myeloma within 6 to 8 weeks before enrolment. Plasmapheresis must not be applied within 2 weeks before enrolment
* Patients with peripheral neuropathy or neuropathic pain of Grade 2 or greater intensity
* Patients with poorly controlled cardio vascular, vascular, pulmonary, gastro-intestinal, endocrine, neurological, psychiatric, hepatic, renal or metabolic diseases or hematological disorders
* Not have oligosecretory or non-secretory multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H, Germany Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (40):
- Germany (40):
  - Augsburg
  - Berlin
  - Bielefeld
  - Bremerhaven
  - Cologne
  - Darmstadt
  - Donauwörth
  - Dresden
  - Frankfurt
  - Halle
  - Hamburg
  - Hamm
  - Hanover
  - Hildesheim
  - Hof
  - Koblenz
  - Lebach
  - Leer
  - Lübeck
  - Magdeburg
  - Mannheim
  - Moers
  - München
  - Münster
  - Neunkirchen
  - Offenburg
  - Oldenburg
  - Osnabrück
  - Passau
  - Porta Westfalica
  - Ravensburg
  - Rostock
  - Saarbrücken
  - Singen
  - Stuttgart
  - Velbert
  - Weiden
  - Wiesbaden
  - Würselen
  - Würzburg

REFERENCES:
- [Derived] Kropff M, Vogel M, Bisping G, Schlag R, Weide R, Knauf W, Fiechtner H, Kojouharoff G, Kremers S, Berdel WE. Bortezomib and low-dose dexamethasone with or without continuous low-dose oral cyclophosphamide for primary refractory or relapsed multiple myeloma: a randomized phase III study. Ann Hematol. 2017 Nov;96(11):1857-1866. doi: 10.1007/s00277-017-3065-z. Epub 2017 Sep 14. PMID 28905189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 23 December 2008 and 10 January 2013 and recruited patients from 42 study centers in Germany.
Pre-assignment Details: A total of 93 participants were randomly allocated and they received at least 1 dose of study drug and were included in the safety analysis. Of these follow-up data on treatment response was not available for 3 participants, so, they were excluded from the Intent-to-treat (ITT) analysis data set and so, ITT included 90 participants.
Period: Treatment Period
Arm/Group | Vd (Bortezomib + Dexamethasone) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide)
Started | 46 (Number of randomized and treated participants) | 47 (Number of randomized and treated participants)
Intent-to-treat Participants | 43 | 47
Completed | 14 (Participants who completed 8 cycles of treatment) | 15 (Participants who completed 8 cycles of treatment)
Not Completed | 32 | 32
Not completed — Adverse Event | 16 | 15
Not completed — Death | 2 | 0
Not completed — Progressive disease | 1 | 0
Not completed — Complete response | 0 | 1
Not completed — Stable disease | 1 | 2
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Non compliance | 0 | 1
Not completed — Reason not specified | 3 | 4
Not completed — Data not available | 1 | 2
Period: Long Term Follow-up
Arm/Group | Vd (Bortezomib + Dexamethasone) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide)
Started | 26 (Number of participants who entered follow-up phase) | 31 (Number of participants who entered follow-up phase)
Completed | 2 (Number of participants who completed follow-up phase) | 0 (Number of participants who completed follow-up phase)
Not Completed | 24 | 31
Not completed — Death | 0 | 4
Not completed — Other | 0 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Progression/Relapse | 22 | 24

BASELINE CHARACTERISTICS:
Population: Number of Intent-to-treat (ITT) participants were included in Baseline analysis. Out of 93 randomized participants (Vd=46; Vcd=47), follow-up data on treatment response was not available for 3 participants, so, they were excluded from the Intent-to-treat (ITT) analysis data set and so, ITT included 90 participants (Vd=43; Vcd=47).
Groups:
- Total: Total of all reporting groups
Arm/Group | Vd (Bortezomib + Dexamethasone) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide) | Total
Number analyzed (Participants) | 43 | 47 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68 (10) | 71 (7) | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 25 | 26 | 51
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 42 | 47 | 89
  African | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression of Disease
Description: 'Median time to progression of disease is assessed according to International Myeloma Working Group (IMWG) criteria or death from any cause. IMWG criteria: increase of >=25% from lowest level in Serum M-component or (the absolute increase must be >=0.5 gram per deciliter [g/dL]); Urine M component or (the absolute increase must be >=200 milligram per 24 hour. Only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain levels. The absolute increase >10 mg/dL. Bone marrow plasma cell percentage >=10%. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing. Development of hypercalcemia. Participants who died or dropped out due to any reason without progression will be censored with the day of death or drop-out, respectively and who are alive at the end of the study without any progression was censored with the last available date.
Time Frame: From the date of randomization until the disease progression or participant's death from any cause whichever occurred first, as assessed up to 72 weeks after end of treatment visit (ie, 46 days after last dose of study medication)
Population: Intent-to-treat (ITT): Participants who received at least one dose of study medication and in whom the primary efficacy parameter could be assessed at least once under study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vd (Bortezomib + Dexamethasone) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide)
Number analyzed (Participants) | 43 | 47
Months | 12.6 [9.83 to 14.43] | 9.9 [8.60 to 11.40]
Statistical Analysis 1: Comparison: Vd (Bortezomib + Dexamethasone) vs Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide); Null Hypothesis: The (median) time to progression is equal in both treatment groups; Test type: Superiority or Other; p = 0.196, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.43 to 1.19]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as time from randomization to myeloma progression according to International Myeloma Working Group (IMWG) criteria or death from any cause. IMWG criteria: increase of ≥25 percent from lowest response level in Serum M-component and/or (the absolute increase must be ≥0.5 g/dL) Urine M-component and/or (the absolute increase must be ≥200 mg/24 hour. Only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain levels. The absolute increase must be >10 mg/dL. Bone marrow plasma cell percentage: the absolute percent must be ≥10 percent. Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas. Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.65mmol/L) that can be attributed solely to the plasma cell proliferative disorder. PFS included disease progression as well as death.
Time Frame: From the date of randomization until the disease progression or participant's death from any cause whichever occured first, as assessed up to 72 weeks after end of treatment visit (ie, 46 days after last dose of study medication)
Population: Intent-to-treat (ITT): all participants who received at least one dose of study medication and in whom the primary efficacy parameter could be assessed at least once under study medication. Participants without progression and who are still alive at the end of the study or dropped out will be censored with the last available date.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vd (Bortezomib + Dexamethasone) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide)
Number analyzed (Participants) | 43 | 47
Months | 12.6 [9.83 to 14.43] | 9.9 [8.60 to 11.40]
Statistical Analysis 1: Comparison: Vd (Bortezomib + Dexamethasone) vs Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide); Test type: Superiority or Other; p = 0.196, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.43 to 1.19]

3. Secondary Outcome: Overall Survival (OS)
Description: Time interval in months time from randomisation to death from any cause.
Time Frame: From the date of randomization until Month 49
Population: Intent-to-treat (ITT): Participants received at least 1 dose of study medication were included in the ITT analysis set. Participants still alive at the end of the study or dropped out will be censored with the last available date.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vd (Bortezomib + Dexamethasone) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide)
Number analyzed (Participants) | 43 | 47
Months | NA [NA to NA] — The values could not be estimated | 41.50 [24.87 to NA] — The upper limit value could not be estimated
Statistical Analysis 1: Comparison: Vd (Bortezomib + Dexamethasone) vs Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide); Test type: Superiority or Other; p = 0.645, Regression, Cox; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.41 to 1.73]

4. Secondary Outcome: Overall Response Rate (ORR) - International Myeloma Working Group (IMWG) Response Criteria
Description: Percentage of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) is reported in the below table. IMWG criteria- CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow; sCR: CR+Normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescencec; PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90%; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24 hour.
Time Frame: Up to 46 days after last bortezomib dose, or as soon as possible after early discontinuation of study treatment or before start of alternative anti-myeloma therapy
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Vd (Bortezomib + Dexamethasone) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide)
Number analyzed (Participants) | 43 | 47
Percentage of participants | 74.4 [NA to NA] | 70.2
Statistical Analysis 1: Comparison: Vd (Bortezomib + Dexamethasone) vs Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide); Test type: Superiority or Other; p = 0.814, Fisher Exact

ADVERSE EVENTS:
Time Frame: Approximately 5 years
Description: A total of 96 patients were randomly allocated to the 2 treatment arms in the study. 93 patients received at least 1 dose of study drug and were included in the safety analysis. Of these follow-up data on treatment response was not available for 3 patients, so, they were excluded from the Intent-to-treat analysis data set.
Arm/Group | Vd (Bortezomib + Dexamethasone) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide)
Serious Adverse Events (participants affected / at risk) | 15/46 | 14/47
Other Adverse Events (participants affected / at risk) | 43/46 | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vd (Bortezomib + Dexamethasone) (N=46) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide) (N=47)
Pneumonia (Infections and infestations) | 4 (4) | 4 (4)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
IIIrd nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 1 (1)
Pituitary haemorrhage (Endocrine disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vd (Bortezomib + Dexamethasone) (N=46) | Vcd (Bortezomib + Low-dose Dexamethasone + Cyclophosphamide) (N=47)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (87) | 18 (83)
Anaemia (Blood and lymphatic system disorders) | 12 (22) | 6 (10)
Leukopenia (Blood and lymphatic system disorders) | 4 (10) | 7 (12)
Neutropenia (Blood and lymphatic system disorders) | 1 (7) | 1 (4)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 17 (28)
Constipation (Gastrointestinal disorders) | 10 (16) | 13 (16)
Nausea (Gastrointestinal disorders) | 7 (7) | 11 (15)
Vomiting (Gastrointestinal disorders) | 3 (5) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 7 (14) | 9 (16)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4) | 9 (13)
Dizziness (Nervous system disorders) | 7 (8) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 5 (11)
Paraesthesia (Nervous system disorders) | 4 (4) | 5 (5)
Dysgeusia (Nervous system disorders) | 3 (3) | 5 (5)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 4 (4)
Neuralgia (Nervous system disorders) | 3 (3) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 2 (2)
Ageusia (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Hemicephalgia (Nervous system disorders) | 0 (0) | 1 (1)
Hypogeusia (Nervous system disorders) | 0 (0) | 1 (1)
Hyposmia (Nervous system disorders) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 13 (15) | 18 (32)
Oedema peripheral (General disorders) | 7 (7) | 10 (13)
Pyrexia (General disorders) | 3 (4) | 7 (10)
Pain (General disorders) | 4 (5) | 5 (5)
Asthenia (General disorders) | 2 (2) | 1 (1)
Oedema (General disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 1 (1)
Local swelling (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 11 (11)
Herpes zoster (Infections and infestations) | 2 (2) | 4 (7)
Bronchitis (Infections and infestations) | 2 (2) | 6 (6)
Respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Eye infection (Infections and infestations) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infective aneurysm (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary mycosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 2 (5)
Weight decreased (Investigations) | 4 (6) | 0 (0)
C-reactive protein increased (Investigations) | 3 (4) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 1 (1)
Weight increased (Investigations) | 2 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Eastern cooperative oncology group performance status worse (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (11) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 3 (4)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis supeficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 4 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Dyssomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2) | 3 (3)
Visual impairment (Eye disorders) | 1 (1) | 4 (4)
Lacrimation increased (Eye disorders) | 1 (2) | 2 (2)
Colour blindness acquired (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 9 (9)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Strangury (Renal and urinary disorders) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days